CLINICAL TRIAL: NCT05640791
Title: Phase II, Single-arm, Exploratory Study to Evaluate the Safety and Effectiveness of Durvalumab Combined With Chemotherapy Neoadjuvant Therapy of Biliary Tract Cancer
Brief Title: Durvalumab Combined With Chemotherapy Neoadjuvant Therapy of Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20220930
Record Dates: First submitted 2022-11-30; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Resectable Biliary Tract Cancer
MeSH Terms: interventions — Cisplatin; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, cisplatin, nab-paclitaxel, durvalumab (Experimental): Participants receive nab-paclitaxel over 30 minutes, cisplatin over 60 minutes, and gemcitabine over 30 minutes on days 1 and 8; durvalumab over 60 minutes on days 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Participants with stable disease (SD), partial response (PR), or complete response (CR) then undergo standard of care hepatectomy with portal lymphadenectomy.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Durvalumab

INTERVENTIONS:
Drug: Cisplatin — 25mg/m2；d1, 8, 21 d cycle
  Other Names: Cisplatinum
Drug: Gemcitabine — 1000mg/m2；d1, 8, 21 d cycle
  Other Names: Difluorodeoxycytidine hydrochloride
Drug: Nab-paclitaxel — 100mg/m2；d1, 8, 21 d cycle
  Other Names: ABI-007
Drug: Durvalumab — 1000mg；d1, 21 d cycle
  Other Names: MEDI4736

SUMMARY:
This phase II trial studies how well gemcitabine, cisplatin, nab-paclitaxel and durvalumab work before surgery in treating participants with Biliary Tract Cancer. The international multicenter phase III clinical study TOPAZ-1 has confirmed that durvalumab combined with gemcitabine and cisplatin can bring survival benefits to advanced BTC. Drugs used in chemotherapy, such as nab-paclitaxel, cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving combination chemotherapy and Durvalumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed as malignant tumor of biliary tract by pathological diagnosis;
2. Computed tomography (CT) or magnetic resonance imaging (MRI) shall be performed with high-quality cross-sectional imaging, and diagnosed as resectable high-risk biliary malignant tumors, limited to the liver, bile duct and/or regional lymph nodes (at least one of the following criteria must be met) :

   * T-stage ≥ Ib (Ib-IV)
   * Solitary lesion > 5 cm
   * Multifocal tumors or satellite lesions present confined to the same lobe of the liver as the dominant lesion but still technically resectable
   * Presence of major vascular invasion but still technically resectable
   * Suspicious or involved regional lymph nodes (N1)
   * No distant extrahepatic disease (M0)
3. The patient's gender is not limited, and the age is 18-75 years old; Life expectancy>3 months;
4. Within one week of enrollment, the ECOG PS score was 0 or 1;
5. No serious complications, such as hypertension, coronary heart disease and psychiatric history, and no serious allergic history; Non pregnancy and non lactation period;
6. The patient's organ and blood system functions meet the requirements:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Platelet count ≥ 100 × 10^9/L
   * Hemoglobin ≥ 90 g/L
   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase ≤ 2.5 x ULN
   * Albumin ≥ 3g/dL
   * Creatinine ≤ 1.5 x ULN
7. The patient can understand and sign the informed consent form to participate in the trial study; can follow up with good compliance.

Exclusion Criteria:

1. Patients who received PD-1, PD-L1, PD-L2, CTLA-4 inhibitors before enrollment, or patients who directly received another stimulatory or co inhibitory T cell receptor (such as CTLA-4, CD137);
2. Used any other research drugs within 4 weeks before enrollment;
3. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism after hormone replacement therapy); Patients with childhood asthma who have completely alleviated and do not need any intervention or leukorrhea after adulthood can be included, but patients who need medical intervention with bronchodilators cannot be included;
4. With congenital or acquired immune deficiency, such as people infected with human immunodeficiency virus (HIV), active hepatitis B (HBV DNA 500IU/ml), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analytical method) or people with hepatitis B and hepatitis C co infection;
5. Severe infection (such as intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first drug administration, or fever of unknown cause>38.5 ° C occurred during screening/before the first drug administration;
6. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Test drug allergy;
8. Suffering from uncontrollable mental illness;
9. Peripheral neuropathy of grade 2 or above according to CTCAE 4.0. In CTCAE 4.0, grade 2 sensory neuropathy is defined as "moderate symptoms; restriction of activities of daily living (ADL)";
10. Occurrence of serious and/or uncontrollable diseases at the same time may affect participation in the study, such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, diabetes out of control, severe activity, uncontrollable infection after inadequate biliary drainage (such as tumor blocking the bile duct), or mental disease/social condition;
11. Pregnancy (positive pregnancy test) or lactation;
12. Diseases of central nervous system (CNS), except for brain metastasis treated. The treated brain metastatic tumor is defined as confirmed by clinical examination and brain imaging (MRI or CT) during the screening period, and there is no sign of progress or bleeding after treatment, and there is no need for continuous application of dexamethasone. Anticonvulsant drugs (stable dosage) are allowed. The treatment of brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; gamma knife, linear accelerator [LINAC] or equivalent) or a combination deemed appropriate by the treating doctor. Patients with central nervous system metastasis who underwent neurosurgical resection or brain biopsy within 3 months before the first day were excluded;
13. Other cancers in the past (within the past 5 years) or at the same time, excluding non melanoma skin cancer and carcinoma in situ;
14. History of allergy or hypersensitivity to any study drug;
15. Current abuse of alcohol or illicit drugs;
16. Unable or unwilling to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of completion of all preoperative and operative therapy | Up to 9 weeks after study start
  Completion of all therapy rate will be recorded.
Incidence of adverse events | Up to 1 years after study start
  Will be monitored using method of Thall, Simon and Estey, and will be tabulated by the maximum reported Common Terminology Criteria for Adverse Events (CTCAE) grade.

SECONDARY OUTCOMES:
Response rate defined as the percentage of patients who will have complete response (CR), partial response (PR) or stable disease (SD) after the neoadjuvant therapy | Up to 9 weeks after study start
  Will be evaluated according to Response Evaluation Criteria in Solid Tumor (RECIST).
Rate of R0 resection | Up to 9 weeks after study start
  R0 resection is defined as no tumor remains at the cutting edge and no tumor cells remain at the cutting edge under the microscope
Recurrence-free survival (RFS) | Up to 1 years after study start
  RFS is defined as the time between the date of surgery and the date of disease recurrence or death, whichever occurred first. If a patient did not have an event (i.e. disease recurrence or death) by the time of final analysis, patient will be censored at the last disease evaluation time.
Overall survival (OS) | Up to 1 years after study start
  OS is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China